CLINICAL TRIAL: NCT00754897
Title: Feasibility Study for Pediatric NeuroDevelopmental Assessment Study (PANDAS)
Brief Title: Feasibility Study for PANDAS
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Ronald Litman, DO, The Children's Hospital of Philadelphia
Other Study IDs: 2008-06-7001
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Inguinal Hernia; Developmental Delay Disorders
Keywords: Phone Interview; Anesthesia; Siblings; Inguinal Hernia; Neurologic Examination; Developmental Delay Disorders
MeSH Terms: conditions — Hernia, Inguinal; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: We will do a database search to identify children less than 1 year of age that have undergone inguinal hernia surgery during the years of 1999-2007, and children who have had inguinal hernia surgery between the ages of 1 and 3 years during the years 1999-2007.
  We will then do a telephone interview of the parents of these children to determine if there are siblings that are within three years of age and have not have any exposure to anesthetics agents or sedatives before their 3rd birthday.

SUMMARY:
We have been asked to participate in the Pediatric Anesthesia NeuroDevelopmental Assessment Study (PANDAS), which is a study to compare neurocognitive functions in sibling pairs: one of whom had exposure to anesthesia during inguinal hernia surgery before three years of age (exposed) and the other who was not exposed to anesthesia or surgery in the first three years of life (unexposed). A consortium of approximately 6 hospitals is doing this feasibility study to determine if there is an adequate number of subjects for each of the two age groups before the formal study begins.

DETAILED DESCRIPTION:
Feasibility study to obtain information through a telephone interview with parents of eligible children Once we identify the children who were less than one year of age and those between the ages of 1 and 3 that who had inguinal hernia surgery during the years of 1999-2007, we will call the parents to determine if the index patients have siblings. If so, we would also ask if there is a sibling within 3 years of the index patient's age and if they have had no exposure to anesthetics or sedatives before their third birthday. Exclusion criteria for both index patients and siblings would include gestational age at birth of < 36 weeks, any history of hospitalization, including neonatal ICU, a history of CNS, cardiac, or pulmonary diseases requiring medical treatment, or a history of subsequent surgery or exposure of anesthetics or sedatives.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 0 to 1 year.
2. Inguinal hernia surgery between 1/1/1999 and 12/31/2007.
3. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Gestational age < 36 weeks.
2. Any history of hospitalization, including neonatal ICU.
3. A history of CNS, cardiac, or pulmonary diseases requiring medical treatment.
4. History of subsequent surgery or exposure to anesthetics or sedatives at less than 3 years of age.

   -

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 1 year of age that have undergone inguinal hernia surgery during the years of 1999-2007, and children who have had inguinal hernia surgery between the ages of 1 and 3 years during the years 1999-2007.
  We will then do a telephone interview of the parents of these children to determine if there are siblings that are within three years of age and have not had any exposure to anesthetics agents or sedatives before their 3rd birthday.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this feasibility study is to determine if there is an adequate population of sibling pairs at CHOP to warrant participation in a future PANDAS study. | 6-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Litman, DO, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States